CLINICAL TRIAL: NCT00056680
Title: Adult Attachment and Intervention Efficacy With Preterms
Brief Title: Three-Part Program for Parents With Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01HD38982-1A6; 1R01HD038982 (NIH)
Record Dates: First submitted 2003-03-20; First posted 2003-03-24 (Estimated); Last update posted 2007-06-20 (Estimated); Status verified 2007-05

CONDITIONS: Premature Birth
Keywords: Prematurity; low birthweight; parenting; intervention
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Psychoeducational video
Behavioral: Infant massage
Behavioral: Brazelton Neonatal Behavioral Assessment Scale

SUMMARY:
This study evaluated the efficacy of a comprehensive, three-part program for parents of premature infants. This program was designed to improve development in preterm children and includes an educational video, tests to evaluate the child's strengths and abilities, and instruction in infant massage.

DETAILED DESCRIPTION:
Premature birth is a major cause of developmental delay, and cost-effective, replicable methods to promote development in preterm children are needed. Despite the success of first generation interventions, little is understood about why early intervention does not affect all parents and preterms to the same degree.

This study assessed the efficacy of a three-component intervention (psychoeducational video, serial administrations of the Brazelton Neonatal Behavioral Assessment Scale, and parent-administered infant massage) that targets preterm infants and their mothers and fathers. Outcome measures included infant physical, intellectual, and socioemotional development; parental sensitivity; and infant-parent attachment. The project also assessed the role of parental state of mind regarding attachment and parental commitment to the intervention.

Participants in this study were urban African American mothers and fathers of preterm, low birthweight infants admitted to the neonatal intensive care unit. Fathers were eligible for the study if nominated by the child's mother. Participants were randomly assigned to an intervention group or a control group. Both groups were comparable with respect to race, maternal pregnancy history, education, income, presence/absence of partner, infant gestational age, infant small-for-date status, and infant gender.

The intervention group viewed a videotape about preterm infant abilities. Over the course of the study, the intervention group administered infant massage and completed multiple administrations of the Brazelton Neonatal Behavioral Assessment Scale with increasing parental involvement.

The intervention began when infants were 32 to 36 weeks post-conceptual age (PCA) and ended when infants are 52 to 56 weeks PCA. The efficacy of the intervention and the moderating roles of adult attachment and parental commitment to the intervention were evaluated in terms of infant physical, mental, motor, and social development, and parental adjustment and sensitivity to the infant during the first 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Infants born < 37 weeks gestational age
* Mothers 18 years of age or older
* African American

Exclusion Criteria:

* Infants with chromosomal abnormalities or other genetic syndromes
* Mothers with positive postpartum toxicology screens
* Infants destined for foster care

Note: age limits for infants refer to post-conceptual age (not actual age)

Ages: 32 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2001-07; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Anthropometrics (weight, height, head circumference), Bayley Scales of Infant Development, infant behavioral problems and behavioral competencies, maternal sensitivity, infant-parent attachment | collected at 4, 12, and 24 months of infant age

SECONDARY OUTCOMES:
Maternal self-efficacy, parenting stress, perceptions of infant temperament | Collected at 4, 12, and 24 months of infant age

CONTACTS AND LOCATIONS:
Overall Officials: Douglas M. Teti, Ph.D., Principal Investigator — The Pennsylvania State University
Locations (5):
- United States (5):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Maryland Medical Center, Baltimore, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - The Pennsylvania State University, University Park, Pennsylvania

REFERENCES:
- [Result] Teti DM, Hess CR, O'Connell M. Parental perceptions of infant vulnerability in a preterm sample: prediction from maternal adaptation to parenthood during the neonatal period. J Dev Behav Pediatr. 2005 Aug;26(4):283-92. doi: 10.1097/00004703-200508000-00004. PMID 16100501
- [Result] Teti, D. M., & Killeen, L. (in press). The role of parental states of mind in effecting parental commitment to an intervention program for premature infants and their parents. In H. Steele & M. Steele (Eds.), The Adult Attachment Interview in Clinical Context. New York: Guilford Press.
- [Result] Candelaria, MA, O'Connell, MA, & Teti, DM. (2006). Cumulative psychosocial and medical risk as predictors of early infant development and parenting stress in an African-American preterm sample. Journal of Applied Developmental Psychology, 27(6), 588-597.